CLINICAL TRIAL: NCT05139823
Title: Extended Cross-sectoral Nurse Follow-up After Discharge From a Geriatric Ward - Benefits and Challenges. A Mixed-method Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karen Andersen-Ranberg, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21/57714
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Extended Cross-sectoral Nurse Follow-up After Discharge From a Geriatric Ward

STUDY DESIGN:
Intervention Model Description: Single-centre two-arm parallel group randomised controlled trial using permuted block randomisation
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization occurs at the time of discharge, meaning that the treatment and post-discharge treatment recommendations given in the ward will not in any way be affected by whether or not the patient is allocated to intervention or control group. Thus, everyone at the geriatric ward is blinded, including the patient, the doctors, nurses, and the investigator who carries out the randomization.
  At discharge the patient is informed about the allocation group. If control, i.e., usual care, nothing further is done. If intervention, the patient, the investigator and the visiting geriatric nurses are made aware of the result of the allocation.
  The outcome assessor is also the investigator, however the results are scrambled by a third party and any identifying information is removed, thus allowing blinded data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Controls receive usual care, which is a digital communication to the local home care team including a discharge care plan to the home care system, including information about the discharge diagnoses, and recommendations for particular attention to specific bodily functions and medical treatment regime. The patient's PCP receives a discharge summary from the treating hospital physician as usual.
- Intervention (Experimental): An appointment for a geriatric follow-up home visit is made with the patient and the municipal home care (community) nurse 2-5 days after discharge and only on weekdays. Relatives are informed about the visit and are welcome to join with the patient's acceptance. The local home care team as well as the patient's PCP receives the same digital discharge plan and discharge summary, respectively, as in the control group. While a follow-up visit is scheduled with the home care nurse, the PCP is invited to join too if available, either in person or by a video link. Administratively, the patients are treated as geriatric outpatients, with an in-home follow up instead of a visit in the Geriatric outpatient clinic.
  Interventions: Procedure: geriatric follow-up home visit after discharge

INTERVENTIONS:
Procedure: geriatric follow-up home visit after discharge — An appointment for a geriatric follow-up home visit is made with the patient and the municipal home care (community) nurse 2-4 days after discharge and only on weekdays. Relatives are informed about the visit and are welcome to join with the patient's acceptance. The local home care team as well as the patient's PCP receives the same digital discharge plan and discharge summary, respectively, as in the control group. While a follow-up visit is scheduled with the home care nurse, the PCP is invited to join too if available, either in person or by a video link. Administratively, the patients are treated as geriatric outpatients, with an in-home follow up instead of a visit in the Geriatric outpatient clinic.
  Arms: Intervention

SUMMARY:
Purpose By using both quantitative and qualitative research methods to examine the impact of a coordinated home visit by a geriatric nurse and a community (home care) nurse to vulnerable older patients recently discharged from a geriatric department. The project will address the transition between health care sectors by examining how nursing care information is communicated between sectors, and whether in-home use of digital health solutions can optimize clinical assessments leading to relevant changes in treatment plans and prevention of acute readmissions. User perspectives of both health professionals, patients and their relatives will be applied.

In the quantitative study the primary endpoints are acute readmissions within 30-days and 90-days. The secondary endpoints are 1 year-mortality, numbers of quantitative clinical assessments (e.g., clinical assessment scores, vital signs, POCT) and their associations with clinical decision making, time to readmission, days out of hospital. Financial costs will be assessed.

The qualitative study will provide insight into the challenges and barriers in the transition between hospital and home and opposite as experienced by the patient. Secondly, with a user perspective (i.e. patient, relatives, health professionals) the study will provide in-depth knowledge in the personal care needs of vulnerable patients and how they can be met in a cross-sectoral collaboration between an out-going geriatric nursing team and the home care nursing team. Finally, the important identified complex areas of nursing care during transition will be described and suggested implemented in educational curricula of health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are patients acutely admitted to G-OUH, residents in Odense Municipality, and discharged to own home with arranged home care for personal care, or discharged to permanent care in a care home.

Exclusion Criteria:

* Excluded from the study are patients discharged to a temporary skilled nursing facility, terminally ill patients with an anticipated short life expectancy, and incapacitated patients, e.g., patients with a diagnosis of dementia or persistent symptoms of cognitive impairment due to delirium during the whole in-hospital stay. Patients with a permanent address in a care home are not excluded by their type of residence unless they are mentally incapacitated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1514 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-12-07 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Acute readmissions | 30 days
  Unplanned readmission within 30 days

SECONDARY OUTCOMES:
Readmission | 90 day
  Unplanned readmission within 90 days
Mortality | 1 year
  1-year mortality
Time to readmission | 1 year
  Hazard model of readmission with a duration of one year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eriksen AV, Beck SH, Nielsen D, Thomsen K, Krone JO, Andersen-Ranberg K. Cross-sectoral follow-up after hospital discharge from a geriatric ward: a study protocol of a randomised controlled trial (G-UD). Trials. 2025 Jul 1;26(1):234. doi: 10.1186/s13063-025-08922-7. PMID 40598384